CLINICAL TRIAL: NCT05182411
Title: Validity and Reliability of Turkish Version Leg Activity Measure
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Zekiye İpek KATIRCI KIRMACI, Asst. Prof., Kahramanmaras Sutcu Imam University
Other Study IDs: ipekkkirmaci
Record Dates: First submitted 2021-12-15; First posted 2022-01-10 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Spinal Cord Injuries; Multiple Sclerosis; Stroke
Keywords: activity; participation; spasticity; passive function; active function
MeSH Terms: conditions — Spinal Cord Injuries; Multiple Sclerosis; Stroke; Motor Activity; Muscle Spasticity | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with spasticity: adult neurological patients with spasticities in their lower extremities
  Interventions: Other: assessment

INTERVENTIONS:
Other: assessment — Turkish version of Leg Activity Measure Rivearmead Mobility Index Nottingham Health Profile Functional Independence Measures

SUMMARY:
Patient-filled scales minimize the burden of data collection for clinicians in a clinical setting.

Therefore, Leg activity measure, a new self-report measure of active and passive function in the leg, has been developed.

Leg activity measure consists of three parts. The first part includes passive functions, the second part includes active functions, and the third part includes the assessment of quality of life.

It is a valid and reliable test in adult neurological patients with lower extremity spasticity. It can be used in the evaluation of the active and passive functions of the results of the clinicians' interventions by making the cultural adaptation of the Turkish language and examining its validity and reliability. We think that it will be important to determine the limitations in activity, participation and daily living activities and to evaluate their reflections.

DETAILED DESCRIPTION:
Spasticity is a common symptom resulting from stroke, brain trauma, and degenerative brain diseases. Spasticity, known as rate-dependent resistance to passive movement, prevents many activities of daily living. Lower extremity spasticity, on the other hand, hinders joint movements and complicates mobility, transfer and passive activities of caregivers.

Goals for the treatment of spasticity often focus on active function improvements in walking, standing, and moving from different sitting positions. However, improvements in passive function tasks and symptom management are often equally important to patients. Active function is the use of the limb to directly perform a task. Passive fonskyion is care of the affected extremity, usually performed by the person himself, but may require assistance from another person.

There is a need for instruments with demonstrable measurement properties that can reflect a clinically significant change in practice. Outcomes developed for treatments such as botulinum toxin and physical interventions for spasticity aimed at improving any aspect of functional performance (active and passive function) should ideally reflect real-life function as opposed to simply observed tasks in the clinical setting.

Leg activity measure filled by the patient consists of three parts. The first part includes passive functions, the second part includes active functions, and the third part includes the assessment of quality of life.

It is a valid and reliable test in adult neurological patients with lower extremity spasticity. It can be used in the evaluation of the active and passive functions of the results of the clinicians' interventions by making the cultural adaptation of the Turkish language and examining its validity and reliability.

ELIGIBILITY:
Inclusion Criteria:

* 1 or more spasticity in at least one muscle according to the Modified Ashworth Scale
* Be between the ages of 18-65
* Volunteering to participate in the study

Exclusion Criteria:

* Under 18 years old, over 65 years old
* History of trauma in the last 1 year
* Having alcohol and substance abuse
* Having a pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult neurological patients with spasticity of the lower extremities
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Turkish version of Leg Activity Measure | First day
  Leg activity measure consists of three parts. The first part includes passive functions, the second part includes active functions, and the third part includes the assessment of quality of life. The questions in each section are scored between 0-4. An increase in the score indicates that the activity could not be performed.
Turkish version of Leg Activity Measure | 2 weeks later
  Leg activity measure consists of three parts. The first part includes passive functions, the second part includes active functions, and the third part includes the assessment of quality of life. The questions in each section are scored between 0-4. An increase in the score indicates that the activity could not be performed.

SECONDARY OUTCOMES:
The Rivermead Mobility Index | First day
  The Rivermead Mobility Index is appropriate for a range of disabilities that include anything from being bedridden to being able to run
Nottingham Health Profile (NHP) | First day
  The NHP is a patient-reported questionnaire. Respondents tick yes or no boxes to answer questions about their health and its effects on their daily life.
  The questionnaire is divided into two parts. The first parts comprises 38 questions in six categories: sleep, physical mobility, energy, pain, emotional reactions, and social isolation.
  The second part of the NHP is made up of seven statements about areas of life that are commonly affected by health: paid employment, jobs around the house, social life, personal relationships, sex life, hobbies and interests, and holidays
The Functional Independence Measure (FIM) | First day
  The Functional Independence Measure (FIM) is an instrument that was developed as a measure of disability for a variety of populations and is not specific to any diagnosis. The FIM instrument includes measures of independence for self-care, including sphincter control, transfers, locomotion, communication, and social cognition.
  Each item is scored on a 7 point ordinal scale, ranging from a score of 1 to a score of 7. The higher the score, the more independent the patient is in performing the task associated with that item.

CONTACTS AND LOCATIONS:
Overall Officials: Zekiye İpek Katırcı Kırmacı, Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaraş Sutcu Imam University, Kahramanmaraş, Turkey (Türkiye)

REFERENCES:
- [Derived] Kirmaci ZIK, Adiguzel H, Kirmaci YS, Tasvuran Horata E, Tuncel Berktas D, Erel S. Turkish translation and transcultural validity and reliability of an assessment tool for spasticity: Leg Activity Measure (Leg A). Neurol Res. 2024 Jul;46(7):644-652. doi: 10.1080/01616412.2024.2340878. Epub 2024 May 2. PMID 38695372